CLINICAL TRIAL: NCT05779228
Title: Visual Mode Switching in Color Perception
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant was not funded
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002354
Record Dates: First submitted 2023-01-20; First posted 2023-03-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Perception of Things Changing Color; Adaptive Behavior
Keywords: Visual Perception; Visual Adaptation; Color Perception

STUDY DESIGN:
Intervention Model Description: The interventional study type is correct. The investigative team is giving all subjects a treatment- behavioral training in visual mode switching- and measuring effects of that treatment, by comparing measures made before to measures made after the treatment. Thus, this is a within-subjects, repeated measures experimental design. The experimenters have 6 different measurements they are using this design in different groups of subjects run in parallel, all examining different effects of the same treatment. . This is why parallel study model is appropriate. These parallel groups with different measurements, but same treatment, are the arms of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Color Contrast (Experimental): Test patch is surrounded spatially by different colors
  Interventions: Behavioral: Mode Switching Training
- Color Adaptation (Experimental): Test patch is surrounded temporally (preceded) by different colors
  Interventions: Behavioral: Mode Switching Training
- Neuroimaging (Experimental): Functional MRI and Electroencephelography data are acquired for multiple test colors
  Interventions: Behavioral: Mode Switching Training
- Red Room (Experimental): Participants are tested in a red-illuminated room
  Interventions: Behavioral: Mode Switching Training
- Dark Room (Experimental): Participants are tested in a completely darkened room
  Interventions: Behavioral: Mode Switching Training
- Gradual Change (Experimental): Participants view a gradual change in tint, presented on a head-mounted display
  Interventions: Behavioral: Mode Switching Training

INTERVENTIONS:
Behavioral: Mode Switching Training — Wear of colored lenses for 1 hr, 5 times per day, for 5 days

SUMMARY:
Participants will be given experience wearing colored lenses that add a tint to the environment. Changes in visual perception and neural processing that arise as a result of this experience will be measured. These are expected as participants learn to switch to "colored lenses mode" where the effects of the lenses are discounted and colors appear more normal as soon as the lenses are put on.

DETAILED DESCRIPTION:
All participants will wear tinted lenses for 1 hour at a time, 5 times per day. Perception (behavior) and neural function (with functional MRI and EEG) before and after this experience will be measured. In the neural measurements, activity will be recorded while participants view stripes of many different colors both with the lenses on and off. In the perceptual measurements, participants will adjust the color of a small patch to appear neutral, neither red nor green. Behavior will be measured in a variety of conditions to test different hypotheses about the origins of the mode-switching effects. These include: 1) surrounding the patch with different colors, 2) preceding the presentation of the patch with presentation of different colors, 3) presenting the tests in a red-illuminated room, 4) presenting the tests in a completely darkened room, and 5) using a head-mount-display (virtual reality goggles) to present simulated lenses that gradually change in strength.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected to normal vision by contact lenses
* No known visual disorders
* Little to no experience in tinted environments (e.g. dark rooms, swimming goggles)

Exclusion Criteria:

* Abnormal color vision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-02-04 (Estimated); Study Completion 2032-02-04 (Estimated)

PRIMARY OUTCOMES:
Change in unique yellow settings | Change will be assessed over the entire study, by comparing a pre-test the day before the intevention (which lasts 5 days) to a post-test the day after the intervention.
  This is a standard psychophysical measure referenced in 100s of papers. Participants adjust a patch of color until it appears neither red nor green and this color is reported in standard colorimetric coordinates (e.g. CIE).
Change in BOLD functional MRI activity | Change will be assessed over the entire study, by comparing a pre-test the day before the intevention (which lasts 5 days) to a post-test the day after the intervention.
  Neural activation will be measured with functional MRI which will be used to measure BOLD activity with standard methods, and reported as percent change from rest, a standard measure, for each voxel in the brain.
Change in EEG activity | Change will be assessed over the entire study, by comparing a pre-test the day before the intevention (which lasts 5 days) to a post-test the day after the intervention.
  Neural activity will be measured with electroencephelography using standard techniques and will be reported as voltage changes over time for each electrode in a standard configuration.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Completely deidentified data, meta-data, stimulus presentation code, and analysis code will be shared following an NIH data sharing plan. Data will be shared using the OSF platform, as well as github for code.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available for at least 10 years, starting at publication date or end of the study.
Access Criteria: Publicly accessible
URL: http://osf.io

REFERENCES:
- [Result] Li Y, Tregillus KE, Luo Q, Engel SA. Visual mode switching learned through repeated adaptation to color. Elife. 2020 Dec 15;9:e61179. doi: 10.7554/eLife.61179. PMID 33320093